CLINICAL TRIAL: NCT01751854
Title: Enhanced Motor Recovery Using Serotonergic Agents in Stroke
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, T. George Hornby, Research Assistant Professor, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU00014257; 1250--018 (Other Grant/Funding Number: NIDRR/FIP - H133G060124)
Record Dates: First submitted 2012-12-14; First posted 2012-12-18 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2012-12

CONDITIONS: Patients With Chronic Stroke
Keywords: pharmacology; rehabilitation; locomotion
MeSH Terms: interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SSRI (Experimental): SSRI alone or with training
  Interventions: Drug: SSRI
- Placebo (Placebo Comparator): Placebo alone or with training
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SSRI — SSRI alone or with training
  Other Names: escitalopram
  Arms: SSRI
Drug: Placebo — Placebo alone or with training
  Arms: Placebo

SUMMARY:
The information derived from this study will be critical to establishing appropriate rehabilitative interventions post-stroke. In particular, traditional use of pharmacological agents to alter motor function post-stroke is directed primarily at reducing the "positive" signs following upper motor neuron lesion, in particular spasticity, or enhanced, velocity-dependent stretch reflex responses to imposed stretch. While pharmacological management of spasticity certainly suppresses clinical and quantitative measures of hypertonia, there is little improvement in functional performance. In contrast, preliminary data on the administration of 5HT agents following neurological injury indicates an increase in motor performance (Pariente 2001) and recovery (Dam 1996), despite an increase in spastic motor activity (Stolp-Smith 1999; see Preliminary Data below). Understanding methods to maximize function following stroke despite potential, short-term increases in spastic motor activity may improve therapeutic intervention strategies. The general objective of this study is therefore to:

1. quantify the effects of short-term SSRI administration on voluntary and spastic motor behaviors in individuals with chronic spastic hemiparesis,
2. identify the changes in impairments and functional recovery of walking ability during BWSTT with the presence or absence of SSRIs.

DETAILED DESCRIPTION:
Walking ability post-stroke is characterized primarily by reduced walking speed and endurance and impaired postural stability which limits functional and societal reintegration. Decreased over ground walking speed is a result of decreased cadence, decreased stride length and increased non-paretic single limb stance duration. Mechanisms underlying reduced velocity are thought to include weakness in the paretic limb, particular hip flexor and plantarflexor strength, but may also be linked spastic motor behaviors and loss of inter- and intra-limb coordination. Rehabilitation efforts to improve strength and muscle coordination patterns during hemiparetic gait may improve gait quality and velocity and therefore improve performance of activities of daily living.

To improve gait performance and functional outcomes following neurological injury, rehabilitation efforts have focused on re-establishing normal walking patterns . Towards this end, the use of body-weight supported treadmill training (BWSTT) has demonstrated significant improvement in walking capability in individuals post-stroke and spinal cord injury . By supporting a portion of a subject's body weight over a treadmill and providing manual facilitation from therapists, previous research has demonstrated improvements in temporal-spatial gait patterns, including gait velocity , endurance (Macko 2005), balance , and symmetry. Importantly, the changes in impairments and functional limitations observed with intensive BWSTT are often greater than that achieved during conventional or lower intensity physical therapy. Given these benefits, particularly in those who require substantial walking assistance following stroke various robotic locomotor retraining devices have been developed to facilitate practice of "kinematically correct" stepping patterns to improve the consistency and duration of treadmill training.

While the changes observed following BWSTT are statistically and functionally significant, it remains unclear is the benefits of such intensive training paradigms are optimized. Specifically, across many larger studies in subjects with chronic stroke (i.e., those > 6 mo. post-injury), mean increases in walking speed range between 0.09 m/s to 0.15 m/s following 1-6 mos. of training. Even in current trials investigating changes in over ground walking speed in robotic- vs. therapist-assisted BWSTT, mean improvements over at least 18 subjects in each group vary from 0.07 to 0.13 m/s, respectively (please see Preliminary work: Pilot Study 1). While again statistically significant, such changes represent an approximate 10% improvement in gait speed as compared to healthy adults (Perry 1992).

To enhance the benefits of intensive BWSTT, many investigators continue to search for combined interventions to augment recovery. One potential adjunct that has received attention is the use of pharmacological agents. For example, anti-spastic medications (e.g., benzodiazepine, baclofen, tizanidine) have been used for decades (to reduce the presence or severity of involuntary, spastic reflexes in patients with stroke. Spasticity has traditionally been thought to be a primary limitation to functional mobility post-stroke, although this premise has been questioned recently . Indeed, many pharmacological agents are effective in reducing spastic motor behaviors although evidence for improvements in function following use of these agents post-stroke is limited. In addition, some evidence suggests that these agents reduce maximal voluntary strength and can impair learning of motor tasks.

New evidence has emerged of a potentially powerful role of excitatory or facilitative modulatory agents in the treatment of motor impairments post-stroke. Based primarily on evidence from experimentally induced lesions in mammals, the application of monoaminergic (i.e., serotonin [5HT] and norepinephrine [NE]) agents excite vs. depress spinal or cortical excitability have gained momentum. In individuals post-stroke, for example, the use of amphetamines (directed primarily through NE pathways) had generated substantial interest as an adjunct to physical therapy interventions, although recent data may suggest no benefit from this agent. Further, the use of amphetamines may enhance the risk of cerebral or coronary vascular disease, which is already compromised in this patient population, and therefore limit the use of these agents in clinical practice.

In contrast, 5HT agents have also been shown to enhance spinal and/or cortical excitability, and may accelerate locomotor recovery following neurological injury when appropriate physical interventions are provided . In humans post-stroke, one study has demonstrated enhanced motor performance and cortical activity following a single dose of SSRIs. In another study of sub-acute stroke, SSRIs and not selective NE reuptake inhibitors improved function during inpatient rehabilitation. Interestingly, a small case report indicates a strong increase in spasticity following use of 5HTergic anti-depressive agents, indicating that both spinal and cortical excitability may contribute to altered motor function. Such findings have been replicated here (please see Preliminary work: Pilot Study I, although certainly require further assessment.

While the above findings are preliminary, two important questions arise. First, if both spastic and voluntary lower extremity activity are simultaneously altered following administration of commonly used anti-depressive medications, how does the relation between these variable alter motor function? Echoing tothers, how important is the prevalence of spasticity to impaired motor function post-stroke? Secondly, can the increased excitability of both spinal and cortical systems following SSRI accelerate motor recovery and the effectiveness of intensive physical rehabilitation strategies, as shown in reduced preparations? Such data are important for health care professionals treating individuals with neurological injury to: A) understand the previously unknown modulation in reflex or voluntary function following a seemingly innocuous agent; and, to B) provide the optimal neural excitability to accelerate motor performance and recovery post-injury.

ELIGIBILITY:
Inclusion Criteria:

* unilateral supratentorial stroke
* MMSE > 22
* > 6 months stroke duration
* < 0.9 m/s gait speed overground

Exclusion Criteria:

* lower extremity contracture
* osteoporosis
* Cardiovascular/metabolic/respiratory instability
* previous central/peripheral nerve injury
* concurrent medications interacting with SSRIs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-12; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Peak treadmill speed | 4 weeks

SECONDARY OUTCOMES:
overground walking speed | 4 weeks

OTHER OUTCOMES:
gait kinematics | 4 weeks
EMG activity | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thomas G Hornby, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Rehabilitation Institute of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Gourab K, Schmit BD, Hornby TG. Increased Lower Limb Spasticity but Not Strength or Function Following a Single-Dose Serotonin Reuptake Inhibitor in Chronic Stroke. Arch Phys Med Rehabil. 2015 Dec;96(12):2112-9. doi: 10.1016/j.apmr.2015.08.431. Epub 2015 Sep 14. PMID 26376447